CLINICAL TRIAL: NCT04007770
Title: Cancer-related Cognitive Function Acupuncture Pilot Study (CLARITY
Brief Title: Acupuncture Pilot Study for Cancer-related Cognitive Function
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 19-179
Record Dates: First submitted 2019-07-02; First posted 2019-07-05 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Stage I Breast Cancer; Stage II Breast Cancer; Stage III Breast Cancer; Stage I Colorectal Cancer; Stage II Colorectal Cancer; Stage III Colorectal Cancer; Gynecologic Cancer; Stage I Gynecologic Cancer; Stage II Gynecologic Cancer; Stage III Gynecologic Cancer; Stage I Prostate Cancer; Stage II Prostate Cancer; Stage III Prostate Cancer
Keywords: Breast Cancer; Colorectal Cancer; Gynecologic Cancer; Acupuncture; Memorial Sloan Kettering Cancer Center; 19-179; Prostate Cancer
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms; Prostatic Neoplasms | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Acupuncture (Experimental)
  Interventions: Other: Acupuncture
- Sham Acupuncture (SA) (Sham Comparator)
  Interventions: Other: Sham Acupuncture
- Wait-List Control (Other): This arm is Closed to accrual.
  Interventions: Other: 16 week waiting period + optional Acupuncture

INTERVENTIONS:
Other: Acupuncture — 10 treatments of acupuncture over the course of 10 weeks with a +/- 7 day window
  Arms: Acupuncture
Other: Sham Acupuncture — 10 treatments of sham acupuncture over the course of 10 weeks with a +/- 7 day window. After the 16-week study concludes patients in this group will have the option of receiving up to 10 sessions of real acupuncture; however, these sessions must be completed within 6 months of study conclusion.
  Arms: Sham Acupuncture (SA)
Other: 16 week waiting period + optional Acupuncture — Optional real acupuncture after 16 weeks waiting period. This arm is Closed to accrual.
  Arms: Wait-List Control

SUMMARY:
This study is being done to explore whether acupuncture can improve cognitive difficulties in patients diagnosed with cancer.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* Age 18 ≥ years old
* Diagnosis (breast, colorectal, prostate or gynecological cancer)
* Completed initial cancer treatment (surgery, chemotherapy, and/or radiation therapy) at least one month prior to study enrollment (patients receiving maintenance cancer treatment with hormonal or targeted therapies are permitted)
* Must report moderate or greater perceived CD as indicated by a score of "quite a bit" or "very much" on at least one of the two items that specifically assess concentration (item #20) and memory (item #25) on the EORTC QLQ-C30 instrument (version 3.0)
* Must indicate that their cognitive functions have worsened since their cancer diagnosis by replying "Yes" to all of the following questions:

  * Do you think or feel that your memory or mental ability has gotten worse since your cancer diagnosis?
  * Do you think your mind isn't as sharp now as it was before your cancer diagnosis?
  * Do you feel like these problems have made it harder to function on your job or take care of things around the home?
* Must be willing to adhere to all study-related procedures, including randomization to one of the 2 possible choices: acupuncture or sham acupuncture

Exclusion Criteria:

* Active disease
* Use of acupuncture for cognitive symptom management within the past 3 months
* Diagnosis of Alzheimer's disease, vascular dementia, Parkinson disease, or other organic brain disorder
* Score of ≥10 on the Blessed Orientation-Memory-Concentration (BOMC) screening instrument
* Primary psychiatric disorder not in remission
* Initiation or change in medication (e.g., hypnotics, sedatives, and/or antidepressants) in the past 8 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Cognitive difficulties as measured by the Functional Assessment of Cancer Therapy - Cognitive Function (FACT-Cog) | 16 weeks
  The perceived cognitive difficulties subscale score of the Functional Assessment of Cancer / FACT-Cog will be the primary outcome for the study.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Mao, MD, MSCE, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (6):
- United States (6):
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org